CLINICAL TRIAL: NCT06076317
Title: Randomized Multicenter Clinical Trial of the Efficacy of a Telemedicine Monitoring in the Management of a Depressive Episode After an Hospitalisation in Medicine or Surgery
Brief Title: Relevance of a Telemedicine Monitoring in the Management of Depression
Acronym: TELEDEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP210990; 2023-A00119-36 (Other: ANSM)
Record Dates: First submitted 2023-07-24; First posted 2023-10-10 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Major Depressive Disorder
Keywords: Characterized depressive disorder; Telemedicine session
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard arm (No Intervention): Patients will have the usual care
- Interventional arm (Experimental): Patients will have telemedicine session
  Interventions: Behavioral: Telemedicine session

INTERVENTIONS:
Behavioral: Telemedicine session — The content of telemedicine session is semi-standardized and includes: (1) evaluation of the tolerance and efficacy of drug treatment; (2) evaluation of depressive symptoms (PHQ9 scale); (3) identification of the daily difficulties; (4 ) personalized advice and orientation towards appropriate care pathways. Among the personalized advice, investigators will use the digital tools available to maintain remission, psychoeducation and monitoring tools (for example, application to learn mindfulness meditation, conversational chatbot coupled with artificial intelligence, etc.). Support on the use of these tools can be provided during telemedicine sessions.
  Arms: Interventional arm

SUMMARY:
Major depressive disorder (MDD) is a common chronic disease. It is the main cause of morbidity and disability in the world with, among other things, an increase in cardio-metabolic risk and a reduction in life expectancy, regardless of suicide risk. MDD is the most expensive medical condition: 10-20 billion €/year in France. This cost is mainly attributable to the functional consequences of the disease, highlighting the medico-economic challenge represented by the optimization of the organization of care.

In France, more than 80% of MDD patients are enrolled in non-psychiatric care pathways, mainly primary care or MSO hospital care (medicine, surgery, obstetrics). Unfortunately, less than half of patients benefit from treatment at an appropriate dosage or duration, thus exposing them to the risks of relapse, recurrence and chronic evolution. It is necessary to optimize this management, in particular by improving secondary prevention, which consists of maintaining treatment in the months following symptomatic remission.

Several support programs (monitoring with assessment of symptomatology) have shown their effectiveness on depressive symptomatology with a favorable medico-economic report, in particular by allowing maintenance of antidepressant treatment. None of these studies have been conducted on French care pathways.

Investigators propose to evaluate the efficacy of telemedicine management (added to usual care) in non-psychiatric care pathways on the evolution of depressive symptomatology for MDD patients. Investigators hypothesize that telemedicine monitoring downstream of MSO hospitalization will increase the response rate to antidepressants at 6 months and reduce the costs attributed to depressive symptoms compared to usual care, in particular by optimizing secondary prevention strategies by maintaining treatment.

The main objective of the research is to assess the efficacy of telemedicine monitoring on depressive symptoms and treatments, added to the out-of-hospital downstream care pathways for patients initially hospitalized in MSO (medicine-surgery-obstetrics), compared to usual care.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a common and often chronic disease. It is the main cause of morbidity and disability in the world with, among other things, an increase in cardio-metabolic risk (diabetes, cardiovascular diseases, high blood pressure) and a reduction in life expectancy, regardless of suicide risk. MDD is the most expensive medical condition: 10-20 billion €/year in France. This cost is mainly attributable to the functional consequences of the disease, highlighting the medico-economic challenge represented by the optimization of the organization of care.

In France, more than 80% of MDD patients are enrolled in non-psychiatric care pathways, mainly primary care or MSO hospital care (medicine, surgery, obstetrics). Unfortunately, less than half of patients benefit from treatment at an appropriate dosage or duration, thus exposing them to the risks of relapse, recurrence and chronic evolution. It is necessary to optimize this management, in particular by improving secondary prevention, which consists of maintaining treatment in the months following symptomatic remission.

Several support programs (monitoring with assessment of symptomatology) have shown their effectiveness on depressive symptomatology with a favorable medico-economic report, in particular by allowing maintenance of antidepressant treatment. None of these studies have been conducted on French care pathways.

Investigators propose to evaluate the efficacy of telemedicine management (added to usual care) in non-psychiatric care pathways on the evolution of depressive symptomatology for MDD patients. Investigators hypothesize that telemedicine monitoring downstream of MSO hospitalization will increase the response rate to antidepressants at 6 months and reduce the costs attributed to depressive symptoms compared to usual care, in particular by optimizing secondary prevention strategies by maintaining treatment.

The main objective of the research is to assess the efficacy of telemedicine monitoring on depressive symptoms and treatments, added to the out-of-hospital downstream care pathways for patients initially hospitalized in MSO (medicine-surgery-obstetrics), compared to usual care.

This is a randomized multicenter clinical trial with two parallel arms concerning a population of MDD patients downstream of an MSO hospitalization evaluating the interest of monitoring by telemedicine of the symptoms and treatments, added to out-of-hospital downstream care pathways compared to usual care. One arm consists in usual care and the other one in usual care + telemedicine monitoring. Included patients will be followed for 3 years, the main endpoint will be the clinical efficacy at 6 months from the start of treatment, as the percentage of patients in remission from depressive symptoms (a reduction in the HADS-depression scale score of 50% or more).

Inclusion is made during MCO hospitalization by the liaison psychiatrist. Will be included patients suffering from a MDD with the indication of antidepressant treatment.

The initial psychometric assessment includes the MINI to verify diagnostic criteria for MDD and the HADS to measure the severity of depressive symptoms. The participants are randomized into two groups: "Usual care + tele-monitoring (UC-Plus)" and "Usual care (UC)".

The "UC" group will follow the care prescribed by the liaison psychiatrist during their hospitalization. Each patient will also receive the contact details of his/her medico-psychological center.

The "UC-Plus" group will follow usual care and benefit from telemedicine sessions led by a nurse/psychologist working under the supervision of a psychiatrist. These sessions follow a standardized protocol with 4 evaluations (maximum duration of 20 minutes): (1) evaluation of the tolerance and efficacy of the psychotropic treatment; (2) assessment of depressive symptoms (PHQ-9 scale); (3) identification of daily difficulties; (4) therapeutic orientation and recommendation. A standardized report (score, evolutionary curve, etc.) validated by a psychiatrist will be sent to the patient and his treating physicians (general practitioner, psychiatrist, oncologist, other). The frequency of sessions is defined by the clinical symptomatology:

* Initially: weekly frequency until response to treatment (reduction of PHQ-9 score>50%)
* After response to treatment: variable frequency (weekly to monthly) decided with the patient until remission (score PHQ-9<5)
* After remission: monthly frequency for 6 months, then end of intervention. An increase in the session frequency is possible in the case of relapse or recurrence.

Evaluations at 3, 6, 12, 18, 24, 30 and 36 months, relating to HADS and medico-economic variables, will be carried out in the 2 arms, by telephone blinded to group membership by a technician clinical study. In the event of a high suicide risk, the patient is referred urgently to appropriate care.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Presence of DSM5 criteria for the diagnosis of a characterized depressive episode
* Patient hospitalized in MCO with request for liaison psychiatry opinion whatever the hospitalization modality (full hospitalization, weekday hospitalization or day hospitalization)
* Initiation, change of molecule or modification of a psychotropic treatment (antidepressant or anxiolytic) during MCO hospitalization by the liaison psychiatrist
* Affiliated or entitled to a social security system (except AME)
* Obtaining free, written and informed consent

Exclusion Criteria:

* Severity of the depressive episode incompatible with outpatient care and relevant to an indication for hospitalization in psychiatry
* Patient is part of a psychiatric care program at the time of the selection visit
* Presence of a mood disorder other than CDD
* Reason for MCO hospitalization secondary to psychiatric disorders, in particular suicide attempts
* MCO hospitalization prolonged beyond 3 weeks after initiation, change of molecule or modification of psychotropic treatment dosage
* Psychiatric comorbidities assessed by psychiatrist, in particular addictions (excluding tobacco), delusional disorders, post-traumatic stress disorder, anxiety disorders (excluding GAD)
* High suicidal risk at the screening visit assessed by psychiatrist
* Presence of a non-psychiatric condition with a vital prognosis of less than 3 years
* Contraindications to telemedicine (no internet access, major vision problems, major cognitive problems, marked impulsivity, clinical situation requiring information to be communicated in person, etc.)
* Conditions making consent impossible (major cognitive disorders, etc.)
* Deprived of liberty or under a protective measure (guardianship or under curatorship)
* Pregnant woman
* Refusal of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 836 (Estimated)
Dates: Start 2024-05-27 (Actual); Primary Completion 2026-08-02 (Estimated); Study Completion 2029-02-02 (Estimated)

PRIMARY OUTCOMES:
Treatment response rate at 6 months after inclusion. | At 6 months
  The response to treatment is defined by a decrease of at least 50% in the Hospital Anxiety and Depression Scale (HADS-Depression) score compared to the baseline. The scale contains 14 items and consists of two subscales: anxiety and depression. Each item is rated on a four-point scale. For the depression score, the minimum value is 0 and the maximum value is 21 in such a way that higher scores mean higher depressive symptoms intensity.

SECONDARY OUTCOMES:
Incremental cost-utility ratio over the 3 years of follow-up | At inclusion, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months and 36 months
  Incremental cost-utility ratio will be measured by a compliance questionnaire
Incremental cost-utility ratio over the 3 years of follow-up | A inclusion, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months and 36 months
  Incremental cost-utility ratio will be assessed by missed medical appointments, visits to the emergency room and the number of sick leave days
Quality of life score | A inclusion, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months and 36 months
  Quality of life score will be assessed by the scale EuroQol - 5 Dimensions - 5 Levels (EQ-5D-5L scale)
  This scale comprises 2 parts:
  * a descriptive questionnaire allowing the assessment of 5 dimensions of health state (mobility, self care, usual activities, pain/discomfort, anxiety/depression), each dimension is scored from 1 to 5 (1=no problem, 5=extreme problem). These 5 scores allow to obtain a five-digit code that will be converted to a single summary number (index value), which reflects how good or bad a health state is according to the preferences of the French general population
  * a visual analogue scale from 0 to 100, where the patient has to report how his health is (0 means the worst health you can imagine and 100 means the best health you can imagine)
Quality of life score | At inclusion, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months and 36 months
  Quality of life score will be assessed by the presenteeism scores on the Stanford Presenteeism Scale (SPS). It is a 6-item self-report questionnaire. Each item is scored from 1 (strongly agree) to 5 (strongly disagree); the items 1,3 and 4 are reverse-scored. The minimum score is 6 and the maximum score is 30. The level of presenteeism increased as the SPS score increased.
Number of relapse episodes for the improvement of secondary prevention objective | At inclusion, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months and 36 months
  Relapse is defined by the presence of the diagnostic criteria for a depressive episode within 6 months of obtaining remission. The diagnostic criteria are assessed on the basis of the 9 DSM-5-TR in the event of an increase in the depression score (HADS, Hospital Anxiety and Depression Scale)
Medication compliance and integration into a psychiatric care pathway | At inclusion, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months and 36 months
  A questionnaire of the treatment adherence will be used. This questionnaire comprises 6 questions and each question can be responded by yes or no. The number of positive answers define the level of compliance: 0 yes means a good level of treatment adherence, 1 or 2 yeses means a mild problem of treatment adherence and 3 yeses or more means a bad level of treatment adherence." Please note that this questionnaire has no defined name.
Medication compliance and integration into a psychiatric care pathway | At inclusion, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months and 36 months
  The time between the liaison psychiatry consultation and the first psychiatric consultation out-of-hospital will be measured
Medication compliance and integration into a psychiatric care pathway | At inclusion, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months and 36 months
  The number of psychiatric and psychological consultations will be evaluated
Medication compliance and integration into a psychiatric care pathway | At inclusion, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months and 36 months
  The total duration of psychiatric or psychological follow-up will be measured
Therapeutic efficacy | At 36 months
  The number of patients with a Hospital Anxiety and Depression Scale (HADS-Depression) score ≤ 7. The scale contains 14 items and consists of two subscales : anxiety and depression. Each item is rated on a four-point scale. For the depression score, the minimum value is 0 and the maximum value is 21 in such a way that higher scores mean higher depressive symptoms intensity.
Evaluation of the feasibility and satisfaction of telemedicine tools by patients included in the experimental group | At inclusion, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months and 36 months
  The number of technical incidents suh as connection errors, connection delays will be measured
Evaluation of the feasibility and satisfaction of telemedicine tools by patients included in the experimental group | At inclusion, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months and 36 months
  Feasibility and satisfaction with the telemedicine tool (administered to the experimental group by the nurse/psychologist on the last telemedicine session) are measured by a 10-item questionnaires based on a 5-degree Likert scale. Each item is scored from 1 to 5 (1 corresponding to "strongly disagree" and 5 to "strongly agree"). The minimum score is 10 and the maximum score is 50. The level of feasibility and satisfaction increases as the score increases.
Evaluation of the satisfaction of depression care | At inclusion, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months and 36 months
  Satisfaction of depression care is measured by a 6-item questionnaires based on a 5-degree Likert scale. Each item is scored from 1 to 5 (1 corresponding to "strongly disagree" and 5 to "strongly agree"). The minimum score is 6 and the maximum score is 30. The level of satisfaction increases as the score increases.
Clinical variables associated with drop out of the care program | At inclusion, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months and 36 months
  In order to assess whether some clinical characteristics may contribute to the drop-out of the telemedecine program, the age (measured in years) will be compared between patients who drop out of the telemedecine program versus patients who fully follow the telemedecine program.
Clinical variables associated with drop out of the care program | At inclusion, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months and 36 months
  In order to assess whether some clinical characteristics may contribute to the drop-out of the telemedecine program, the level of education (measured in years spent in education) will be compared between patients who drop out of the telemedecine program versus patients who fully follow the telemedecine program.
Clinical variables associated with drop out of the care program | At inclusion, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months and 36 months
  In order to assess whether some clinical characteristics may contribute to the drop-out of the telemedecine program, the gender (qualitative variable: male - female - other) will be compared between patients who drop out of the telemedecine program versus patients who fully follow the telemedecine program.
Clinical variables associated with drop out of the care program | At inclusion, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months and 36 months
  In order to assess whether some clinical characteristics may contribute to the drop-out of the telemedecine program, the professional status (qualitative variable: in activity - without activity - student - retired) will be compared between patients who drop out of the telemedecine program versus patients who fully follow the telemedecine program.
Clinical variables associated with drop out of the care program | At inclusion, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months and 36 months
  In order to assess whether some clinical characteristics may contribute to the drop-out of the telemedecine program, the marital status (qualitative variable: single - in a relationship - married - divorced - widow) will be compared between patients who drop out of the telemedecine program versus patients who fully follow the telemedecine program.
Clinical variables associated with drop out of the care program | At inclusion, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months and 36 months
  In order to assess whether some clinical characteristics may contribute to the drop-out of the telemedecine program, the main diagnosis (qualitative variable: diagnosis in the International Classification of Diseases ICD-10) will be compared between patients who drop out of the telemedecine program versus patients who fully follow the telemedecine program.
Clinical variables associated with drop out of the care program | At inclusion, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months and 36 months
  In order to assess whether some clinical characteristics may contribute to the drop-out of the telemedecine program, the nature of the psychotic treatment (qualitative variable: benzodiazepin, SSRI antidepressant, tricyclic antidepressant, SNRI antidepressant, typical antipsychotic, atypical antipsychotic, antihistamine drugs, mood stabilizers) will be compared between patients who drop out of the telemedecine program versus patients who fully follow the telemedecine program.
Measurement of stigma scale scores and subscores in each group | At inclusion and 6 months
  Measuring the level of stigma before and after intervention with the Stigma Scale in order to assess the effect of the monitoring on the stigma experienced. The Stigma Scale is a 28-item self-report questionnaire. Each item is scored from 0 (strongly agree) to 4 (strongly disagree). The minimum score is 0 and the maximum score is 112. The level of stigma increased as the score decreased.
Evaluation of the possibility of the physicians to require a psychiatric opinion on the care | At inclusion, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months and 36 months
  Number of telephone calls from physicians to the psychiatrist of the telemedicine platform
Identification of the use of NICT tools (New Information and Communication technologies) | At inclusion, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months and 36 months
  Identification of the NICT (New Information and Communication technologies) used in the field of mental health in each of the groups at each evaluation time (qualitative variable : name of the NICT tool)
Frequency of the use of NICT tools (New Information and Communication technologies) | At inclusion, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months and 36 months
  Frequency of the use of identified NICT (New Information and Communication technologies) used in the field of mental health in each of the groups at each evaluation time (quantitative variable : the reported number of use per week since the last evaluation)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Yves ROTGE, Pr, Principal Investigator — Hôpital Pitié Salpêtrière - Assistance Publique Hôpitaux de Paris
Locations (1):
- Hôpital Pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients. Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.